CLINICAL TRIAL: NCT03119259
Title: Technology Intervention to Support Caregiving for Alzheimer's Disease (I-CARE)
Acronym: I-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Richard Holden, Professor of Health & Wellness Design, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1606267154; R21AG062966 (NIH)
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Dementia, Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC Clinical Program Only and Usual Care (Active Comparator): Patients and informal caregivers randomized to the comparison group will receive care provided by the ABC Clinical Program and IUHP. The ABC Clinical Program is the standard of ADRD care at Eskenazi Health and Primary Care Visits at Indiana University Health is the usual care.
  Interventions: Behavioral: ABC Clinical Program
- BCN Mobile App Plus ABC and BCN Mobile app only (Experimental): Patients and caregivers randomized to the intervention group will continue to receive care in ABC clinical program and IUHP, and have the BCN software installed on either the caregiver's personal mobile device (assuming it meets minimal technical requirements) or a device provided by the study, per participant preference. A research assistant will orient participants to the device, provide training on the BCN software, and troubleshoot technical issues. Participants will receive daytime technical support by phone, electronic support request through a separate app, or printed and in-app help manuals. Hardware, software, and connectivity check-ups will be provided by study research personnel.
  Interventions: Behavioral: ABC Clinical Program; Behavioral: BCN

INTERVENTIONS:
Behavioral: ABC Clinical Program — The goal of the ABC Clinical Program is to help primary care physicians achieve the standard of care in the diagnosis, evaluation and management of patients with ADRD. The ABC Clinical Program is delivered by an interdisciplinary team led by a care coordinator. The informal caregiver is also enrolled in the program and caregiver burden is assessed and managed. The ABC team collects all relevant data and formulates an individualized care plan in collaboration with the informal caregiver. The care coordinator communicates the team's recommendations to the primary care physician and finalizes a collaborative plan of action. During the next year, the ABC team uses face-to-face and telephone interactions with the patient and caregiver to monitor and modify implementation of the care plan.
  The goal of IUHP Usual Care is to provide preventive care services to their patients. Older adults are assessed for ADRD during clinic visits and refered to brain care specialty as necessary.
  Other Names: IUHP Usual Care
Behavioral: BCN — BCN is a mobile application (app) for informal caregivers of patients with Alzheimer's Disease and related dementias (ADRD). The BCN app delivers the following behavioral support:
  1. 24/7 psychoeducation and caregiver support on a variety of ADRD related topics, presented as a browse-able library of stories and advice cards or "Notes";
  2. Assessment of informal caregiver status and patients behavioral and psychological symptoms of dementia (BPSD), in the form of the selfadministered HABC Monitor, along with reporting and historical tracking of HABC Monitor scores;
  3. Engagement tools, in particular, (i) a toolkit for saving, sorting, creating/editing, and sharing Notes and (ii) a bi-directional messaging tool for communicating with clinicians or trusted others.
  Arms: BCN Mobile App Plus ABC and BCN Mobile app only

SUMMARY:
The specific aims of this study are 1) to test the trial and intervention feasibility of Brain Care Notes (BCN) app, 2) To estimate the effect size of BCN on reducing informal caregiver burden at 6 months, and 3) To estimate the effect size of BCN on reducing patient behavioral and psychological symptoms of dementia (BPSD) at 6 months. Subjects will be recruited from the Aging Brain Care (ABC) program of Eskenazi Health and Indiana University Health located in central Indiana.

DETAILED DESCRIPTION:
Informal caregivers of patients with Alzheimer's disease and related dementia (ADRD) manage a complex spectrum of patient behavioral and psychological symptoms of dementia (BPSD). BPSD are major contributing factors to caregivers' burden and adverse health outcomes, leading to an increase of unplanned hospitalizations and a decrease in quality of life. The National Alzheimer's Project Act recognizes the need for interventions that "enable family caregivers to continue to provide care while maintaining their own health and well-being." Furthermore, recommendations from 2015 and 2018 Alzheimer's Disease Research Summits include the application of technology to improve caregiving research and ADRD care

This pilot randomized controlled trial, will test the feasibility and estimate the effect size of integrating mobile health technology BrainCare Notes (BCN) into an existing, fully operational, and self-sustaining clinical program (Aging Brain Care; ABC) and IU Health primary care physician clinics (IUHP). BCN is a mobile application (app) for informal caregivers of patients with Alzheimer's Disease and related dementia (ADRD). The BCN app delivers 24/7 psychoeducation and caregiver support, assessment of informal caregiver status and patients' behavioral and psychological symptoms of dementia (BPSD), and engagement tools for self-management and communication. Over a 15 month accrual period, we propose to enroll from the ABC clinical program and IUHP 60 dyads consisting of an adult patient with ADRD and one (primary) informal caregiver. The intervention will continue for 6 months and final assessments will be completed at 6 months. Feasibility data will be collected throughout the study and assessed at the end of the study by computing: (a) recruitment rate; (b) data completion; (c) BCN usability; (d) BCN acceptance; and (e) BCN use. Caregiver burden and patient BPSD will be collected at baseline, 3, and 6 months and evaluated for changes from baseline to 6 months in each group. Means, standard deviations, and confidence intervals will be computed to test feasibility hypotheses. Mixed linear models will be used to test hypotheses comparing the two conditions at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received a diagnosis of possible or probable Alzheimer's disease and Related Dementia from a physician in the ABC Clinical Program;
* Caregiver is at least 18 years of age and does not have a visual impairment significant enough to interfere with his/her ability to use BCN;
* Both patient and caregiver are community-dwelling in central Indiana; and
* Both patient and caregiver are willing to participate in the ABC Clinical Program (including receiving home visits).

Exclusion Criteria:

* Either the patient or his/her informal caregiver does not have the ability to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Holden, PhD, Principal Investigator — Indiana University; Malaz Boustani, MD, MPH, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Data, or results, will be shared through traditional mechanisms such as peer-reviewed journals and presentations at national meetings. The Enhanced Medical Record - Aging Brain Care (eMR-ABC), the dedicated electronic medical record for the Aging Brain Care (ABC) Clinical Program, was developed with the intent of sharing de-identified data with the scientific community. The Indiana Network for Patient Care (INPC) is a state-wide health information exchange. INPC data is collected for patient care purposes and is not "owned" by Indiana University or the Regenstrief Institute, Inc. - each participating health care system or program retains ownership of their data. At present, Indiana University/Regenstrief Institute scientists do not have the direct authority to share even de-identified patient data. Therefore, any request to use these data for research purposes must be adjudicated on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10 years from the completion of the study
Access Criteria: To obtain IDP, requesters must provide a CV or biosketch detailing their institutional affiliation(s), the scientific purpose for the data sharing request, and plans for the safe and secure management of deidentified study data.

REFERENCES:
- [Derived] Braly T, Muriathiri D, Brown JC, Taylor BM, Boustani MA, Holden RJ. Technology intervention to support caregiving for Alzheimer's disease (I-CARE): study protocol for a randomized controlled pilot trial. Pilot Feasibility Stud. 2021 Jan 11;7(1):23. doi: 10.1186/s40814-020-00755-2. PMID 33431027

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Dyads of informal caregivers plus patients randomized to the comparison group receive usual care for Alzheimer's disease and related dementia (ADRD) from their health system, either Eskenazi Health or Indiana University (IU) Health.
  The standard of ADRD care at Eskenazi Health is the ABC Clinical Program. The goal of the ABC Clinical Program is to help primary care physicians achieve the standard of care in the diagnosis, evaluation and management of patients with ADRD. It is delivered by an interdisciplinary team led by a care coordinator. The informal caregiver of the person living is also enrolled in the program and caregiver burden is assessed and managed. The ABC team collects all relevant data and formulates an individualized care plan in collaboration with the informal caregiver. The care coordinator communicates the team's recommendations to the primary care physician and finalizes a collaborative plan of action. During the next year, the ABC team uses face-to-face and telephone interactions with the patient and caregiver to monitor and modify implementation of the care plan.
  The standard of ADRD care at IU Health is Primary Care visits. The goal of Primary Care at IU Health is to provide preventive care services to their patients. Older adults are assessed for ADRD during clinic visits and referred to brain care specialty as necessary.
- Brain CareNotes (BCN) Software: Dyads of informal caregivers plus patients randomized to the intervention group continue to receive usual care for ADRD at Eskenazi Health or IU Health, and additionally receive the BCN software.
  BCN is installed on either the caregiver's personal mobile device or a device provided by the study. A research assistant orients participants to the device, provides training on the BCN software, and provides technical support and reminders.
  BCN is a mobile application (app) for informal caregivers of patients with ADRD. The BCN app delivers the following behavioral support:
  1. 24/7 psychoeducation and caregiver support on a variety of ADRD related topics, presented as a browse-able library of stories and advice cards or "Notes";
  2. Assessment of informal caregiver status and patients behavioral and psychological symptoms of dementia (BPSD), in the form of the selfadministered HABC Monitor, along with reporting and historical tracking of HABC Monitor scores;
  3. Engagement tools, in particular, (i) a toolkit for saving, sorting, creating/editing, and sharing Notes and (ii) a bi-directional messaging tool for communicating with clinicians or trusted others.
Period: Overall Study
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Started (This table displays number of dyads. Each dyad comprises one patient and their informal caregiver) | 27 | 26
Completed (This table displays number of dyads. Each dyad comprises one patient and their informal caregiver) | 22 | 23
Not Completed | 5 | 3
Not completed — Withdrawn as no longer eligible | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Usual Care (Caregiver Characteristics); Usual Care (Patient Characteristics): Dyads of informal caregivers plus patients randomized to the comparison group receive usual care for Alzheimer's disease and related dementia (ADRD) from their health system, either Eskenazi Health or Indiana University (IU) Health.
  The standard of ADRD care at Eskenazi Health is the ABC Clinical Program. The goal of the ABC Clinical Program is to help primary care physicians achieve the standard of care in the diagnosis, evaluation and management of patients with ADRD. It is delivered by an interdisciplinary team led by a care coordinator. The informal caregiver of the person living is also enrolled in the program and caregiver burden is assessed and managed. The ABC team collects all relevant data and formulates an individualized care plan in collaboration with the informal caregiver. The care coordinator communicates the team's recommendations to the primary care physician and finalizes a collaborative plan of action. During the next year, the ABC team uses face-to-face and telephone interactions with the patient and caregiver to monitor and modify implementation of the care plan.
  The standard of ADRD care at IU Health is Primary Care visits. The goal of Primary Care at IU Health is to provide preventive care services to their patients. Older adults are assessed for ADRD during clinic visits and referred to brain care specialty as necessary.
- Brain CareNotes (BCN) Software (Caregiver Characteristics); Brain CareNotes (BCN) Software (Patient Characteristics): Dyads of informal caregivers plus patients randomized to the intervention group continue to receive usual care for ADRD at Eskenazi Health or IU Health, and additionally receive the BCN software.
  BCN is installed on either the caregiver's personal mobile device or a device provided by the study. A research assistant orients participants to the device, provides training on the BCN software, and provides technical support and reminders.
  BCN is a mobile application (app) for informal caregivers of patients with ADRD. The BCN app delivers the following behavioral support:
  1. 24/7 psychoeducation and caregiver support on a variety of ADRD related topics, presented as a browse-able library of stories and advice cards or "Notes";
  2. Assessment of informal caregiver status and patients behavioral and psychological symptoms of dementia (BPSD), in the form of the selfadministered HABC Monitor, along with reporting and historical tracking of HABC Monitor scores;
  3. Engagement tools, in particular, (i) a toolkit for saving, sorting, creating/editing, and sharing Notes and (ii) a bi-directional messaging tool for communicating with clinicians or trusted others.
- Total: Total of all reporting groups
Arm/Group | Usual Care (Caregiver Characteristics) | Brain CareNotes (BCN) Software (Caregiver Characteristics) | Usual Care (Patient Characteristics) | Brain CareNotes (BCN) Software (Patient Characteristics) | Total
Number analyzed (Participants) | 27 | 26 | 27 | 26 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age unknown for 4 participants
  years
    number analyzed (Participants) | 27 | 26 | 25 | 24 | 102
    (all) | 63.3 (13.0) | 62.5 (13.7) | 77.2 (9.9) | 76.0 (10.6) | 62.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex unknown for 2 participants
  Participants
    number analyzed (Participants) | 27 | 26 | 25 | 26 | 104
    Female | 22 | 19 | 18 | 15 | 74
    Male | 5 | 7 | 7 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 25 | 26 | 25 | 25 | 101
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 12 | 10 | 12 | 46
  White | 14 | 14 | 16 | 13 | 57
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Marital status [Count of Participants; unit: Participants]
  Married | 22 | 16 | 0 | 0 | 38
  Living with partner | 0 | 1 | 0 | 0 | 1
  Divorced | 2 | 2 | 0 | 0 | 4
  Separated | 0 | 1 | 0 | 0 | 1
  Never married | 3 | 6 | 0 | 0 | 9
  Not measured | 0 | 0 | 27 | 26 | 53
Caregiver living situation [Count of Participants; unit: Participants]
  Lives with spouse | 19 | 14 | 0 | 0 | 33
  Lives with children's family | 1 | 2 | 0 | 0 | 3
  Lives with spouse and children's family | 3 | 3 | 0 | 0 | 6
  Lives alone | 1 | 4 | 0 | 0 | 5
  Other | 3 | 3 | 0 | 0 | 6
  Not measured | 0 | 0 | 27 | 26 | 53
Insurance [Count of Participants; unit: Participants]
  Medicare | 2 | 1 | 0 | 0 | 3
  Medicaid | 3 | 2 | 0 | 0 | 5
  Medicare + Medicaid | 1 | 2 | 0 | 0 | 3
  Private/commercial | 7 | 7 | 0 | 0 | 14
  Medicare + Private | 12 | 10 | 0 | 0 | 22
  Self Pay/None | 1 | 2 | 0 | 0 | 3
  Private + Self Pay | 1 | 2 | 0 | 0 | 3
  Not measured | 0 | 0 | 27 | 26 | 53
Employment [Count of Participants; unit: Participants]
  Employed full time (40 hours or more) | 9 | 8 | 0 | 0 | 17
  Employed part time (less than 40 hours) | 0 | 3 | 0 | 0 | 3
  Unemployed | 0 | 2 | 0 | 0 | 2
  Retired | 13 | 12 | 0 | 0 | 25
  Homemaker | 3 | 0 | 0 | 0 | 3
  On social security or disability | 2 | 1 | 0 | 0 | 3
  Not measured | 0 | 0 | 27 | 26 | 53
Income [Count of Participants; unit: Participants]
  $10,000 or less | 0 | 3 | 0 | 0 | 3
  $10,001 to $30,000 | 8 | 7 | 0 | 0 | 15
  $30,001 to $50,000 | 6 | 7 | 0 | 0 | 13
  $50,001 to $75,000 | 4 | 4 | 0 | 0 | 8
  $75,001 to $100,000 | 4 | 2 | 0 | 0 | 6
  $100,001 or above | 4 | 2 | 0 | 0 | 6
  Unknown | 1 | 1 | 0 | 0 | 2
  Not measured | 0 | 0 | 27 | 26 | 53
Education [Count of Participants; unit: Participants]
  Grade School or Middle School | 0 | 0 | 0 | 0 | 0
  Some High School | 3 | 2 | 0 | 0 | 5
  High School Graduate or GED | 6 | 4 | 0 | 0 | 10
  Some College | 4 | 6 | 0 | 0 | 10
  College Degree | 6 | 6 | 0 | 0 | 12
  Masters or other advanced degree | 8 | 8 | 0 | 0 | 16
  Unknown | 0 | 0 | 0 | 0 | 0
  Not measured | 0 | 0 | 27 | 26 | 53
Years caring for person with ADRD [Count of Participants; unit: Participants]
  1 year or less | 4 | 4 | 0 | 0 | 8
  2 years | 3 | 5 | 0 | 0 | 8
  3 years | 7 | 4 | 0 | 0 | 11
  4 years | 3 | 4 | 0 | 0 | 7
  5 years | 4 | 2 | 0 | 0 | 6
  6 years or more | 6 | 7 | 0 | 0 | 13
  Not measured | 0 | 0 | 27 | 26 | 53
Hours per day spent caregiving [Count of Participants; unit: Participants]
  0-1 hours | 1 | 3 | 0 | 0 | 4
  2-5 hours | 3 | 6 | 0 | 0 | 9
  6-9 hours | 8 | 0 | 0 | 0 | 8
  10-13 hours | 5 | 3 | 0 | 0 | 8
  14-17 hours | 3 | 3 | 0 | 0 | 6
  18+ hours | 7 | 11 | 0 | 0 | 18
  Not measured | 0 | 0 | 27 | 26 | 53
Single Item Literacy Screener [Count of Participants; unit: Participants] — Participants were asked to rate their need for help reading heath information on a five-point scale (Never, Rarely, Sometimes, Often, Always)
  Participants
    Never | 19 | 16 | 0 | 0 | 35
    Rarely | 7 | 6 | 0 | 0 | 13
    Sometimes | 1 | 3 | 0 | 0 | 4
    Often | 0 | 1 | 0 | 0 | 1
    Always | 0 | 0 | 0 | 0 | 0
    Not measured | 0 | 0 | 27 | 26 | 53
Study site [Count of Participants; unit: Participants]
  Eskenazi Health | 17 | 16 | 17 | 16 | 66
  IU Health | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Recruitment Rate
Description: Recruitment rate is the average monthly rate of recruitment into the study, calculated as participants recruited over the accrual period.
Time Frame: 15 month accrual period
Population: Caregivers recruited to the study
Measure: Mean (Standard Deviation); unit: participants recruited per month
Groups:
- All Participants: All participants, prior to assignment to condition
Arm/Group | All Participants
Number analyzed (Participants) | 61
participants recruited per month | 4.1 (4.1)

2. Primary Outcome: Feasibility: Data Completeness
Description: Data completeness is the number of enrolled and randomized individuals who provided data at 3 and 6 months.
Time Frame: 6 months after enrollment and randomization
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: Informal caregivers randomized to the comparison group receive usual care for Alzheimer's disease and related dementia (ADRD) from their health system, either Eskenazi Health or Indiana University (IU) Health.
  The standard of ADRD care at Eskenazi Health is the ABC Clinical Program. The goal of the ABC Clinical Program is to help primary care physicians achieve the standard of care in the diagnosis, evaluation and management of patients with ADRD. It is delivered by an interdisciplinary team led by a care coordinator. The informal caregiver of the person living is also enrolled in the program and caregiver burden is assessed and managed. The ABC team collects all relevant data and formulates an individualized care plan in collaboration with the informal caregiver. The care coordinator communicates the team's recommendations to the primary care physician and finalizes a collaborative plan of action. During the next year, the ABC team uses face-to-face and telephone interactions with the patient and caregiver to monitor and modify implementation of the care plan.
  The standard of ADRD care at IU Health is Primary Care visits. The goal of Primary Care at IU Health is to provide preventive care services to their patients. Older adults are assessed for ADRD during clinic visits and referred to brain care specialty as necessary.
- Brain CareNotes (BCN) Software: Informal caregivers randomized to the intervention group continue to receive usual care for ADRD at Eskenazi Health or IU Health, and additionally receive the BCN software.
  BCN is installed on either the caregiver's personal mobile device or a device provided by the study. A research assistant orients participants to the device, provides training on the BCN software, and provides technical support and reminders.
  BCN is a mobile application (app) for informal caregivers of patients with ADRD. The BCN app delivers the following behavioral support:
  1. 24/7 psychoeducation and caregiver support on a variety of ADRD related topics, presented as a browse-able library of stories and advice cards or "Notes";
  2. Assessment of informal caregiver status and patients behavioral and psychological symptoms of dementia (BPSD), in the form of the selfadministered HABC Monitor, along with reporting and historical tracking of HABC Monitor scores;
  3. Engagement tools, in particular, (i) a toolkit for saving, sorting, creating/editing, and sharing Notes and (ii) a bi-directional messaging tool for communicating with clinicians or trusted others.
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
Participants
  3 months | 19 | 21
  6 months | 22 | 23

3. Primary Outcome: Feasibility: BCN Usability (3 Months)
Description: BCN usability at 3 months is the summary score on the modified System Usability Scale (SUS) 10-item scale instrument, ranging from 0 (worst outcome) to 100 (best outcome).
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Brain CareNotes (BCN) Software App: Participants allocated to the BCN app intervention
Arm/Group | Brain CareNotes (BCN) Software App
Number analyzed (Participants) | 20
score on a scale | 76.3 [66.3 to 83.8]

4. Primary Outcome: Feasibility: BCN Usability (6 Months)
Description: BCN usability at 6 months is the summary score on the modified System Usability Scale (SUS) 10-item scale instrument, ranging from 0 to 100. Higher scores indicate higher usability.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Brain CareNotes (BCN) Software App
Number analyzed (Participants) | 21
score on a scale | 72.5 [70 to 90]

5. Primary Outcome: Feasibility: BCN Acceptance (3 Months)
Description: Acceptance at 3 months is the mean score on the Behavioral Intention 4-item scale on a 7-point response scale from 0 (not at all) to 6 (a great deal). Higher scores indicate higher acceptance.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Brain CareNotes (BCN) Software App
Number analyzed (Participants) | 17
score on a scale | 2 [1.5 to 4.0]

6. Primary Outcome: Feasibility: BCN Acceptance (6 Months)
Description: Acceptance at 6 months is the mean score on the Behavioral Intention 4-item scale on a 7-point response scale from 0 (not at all) to 6 (a great deal).
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Brain CareNotes (BCN) Software App
Number analyzed (Participants) | 21
score on a scale | 2.0 [1.0 to 3.0]

7. Secondary Outcome: Caregiver Burden (Baseline)
Description: Informal caregiver burden at baseline, assessed by calculating the NPI-Caregiver Distress score (possible range from 0, best outcome, to 60, worst outcome) from the researcher administered Neuropsychiatric Inventory (NPI)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
score on a scale | 9.8 (7.4) | 8.5 (6.3)

8. Secondary Outcome: Caregiver Burden (3 Months)
Description: Informal caregiver burden at 3 months, assessed by calculating the NPI-Caregiver Distress score (possible range from 0, best outcome, to 60, worst outcome) from the researcher administered Neuropsychiatric Inventory (NPI)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
score on a scale | 10.9 (8.2) | 7.5 (6.8)

9. Secondary Outcome: Caregiver Burden (6 Months)
Description: Informal caregiver burden at 6 months, assessed by calculating the NPI-Caregiver Distress score (possible range from 0, best outcome, to 60, worst outcome) from the researcher administered Neuropsychiatric Inventory (NPI)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
score on a scale | 8.8 (7.0) | 7.8 (6.2)

10. Secondary Outcome: BPSD Severity (Baseline)
Description: Severity of patient behavioral and psychological symptoms of dementia (BPSD) at baseline, assessed by calculating the NPI total score (possible range from 0, best outcome, to 144, worst outcome) from caregiver-reported responses to the researcher-administered Neuropsychiatric Inventory (NPI).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
score on a scale | 17.2 (15.5) | 16.4 (13.4)

11. Secondary Outcome: BPSD Severity (3 Months)
Description: Severity of patient behavioral and psychological symptoms of dementia (BPSD) at 3 months, assessed by calculating the NPI total score (possible range from 0, best outcome, to 144, worst outcome) from caregiver-reported responses to the researcher-administered Neuropsychiatric Inventory (NPI).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
score on a scale | 18.3 (15.1) | 12.4 (11.0)

12. Secondary Outcome: BPSD Severity (6 Months)
Description: Severity of patient behavioral and psychological symptoms of dementia (BPSD) at 6 months, assessed by calculating the NPI total score (possible range from 0, best outcome, to 144, worst outcome) from caregiver-reported responses to the researcher-administered Neuropsychiatric Inventory (NPI).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 27 | 26
score on a scale | 18.5 (16.0) | 15.9 (12.9)

13. Secondary Outcome: Acute Care Utilization (3 Months)
Description: Number of all-cause hospital and emergency room admissions among patients and caregivers in the first 3 months (3 months post-intervention).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 19 | 21
Participants
  Patients | 7 | 13
  Caregivers | 5 | 6

14. Secondary Outcome: Acute Care Utilization (6 Months)
Description: Number of all-cause hospital and emergency room admissions among patients and caregivers in the last 3 months (at 6 months post-intervention).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Brain CareNotes (BCN) Software
Number analyzed (Participants) | 22 | 23
Participants
  Patients | 3 | 13
  Caregivers | 5 | 3

ADVERSE EVENTS:
Time Frame: 6 months from enrollment
Description: Adverse events among caregiver participants were collected and reported separately from patient participants
Groups:
- Usual Care - Caregivers: Informal caregivers randomized to the comparison group receive usual care for Alzheimer's disease and related dementia (ADRD) from their health system, either Eskenazi Health or Indiana University (IU) Health.
  The standard of ADRD care at Eskenazi Health is the ABC Clinical Program. The goal of the ABC Clinical Program is to help primary care physicians achieve the standard of care in the diagnosis, evaluation and management of patients with ADRD. It is delivered by an interdisciplinary team led by a care coordinator. The informal caregiver of the person living is also enrolled in the program and caregiver burden is assessed and managed. The ABC team collects all relevant data and formulates an individualized care plan in collaboration with the informal caregiver. The care coordinator communicates the team's recommendations to the primary care physician and finalizes a collaborative plan of action. During the next year, the ABC team uses face-to-face and telephone interactions with the patient and caregiver to monitor and modify implementation of the care plan.
  The standard of ADRD care at IU Health is Primary Care visits. The goal of Primary Care at IU Health is to provide preventive care services to their patients. Older adults are assessed for ADRD during clinic visits and referred to brain care specialty as necessary.
- Brain CareNotes (BCN) Software - Caregivers: Informal caregivers randomized to the intervention group continue to receive usual care for ADRD at Eskenazi Health or IU Health, and additionally receive the BCN software.
  BCN is installed on either the caregiver's personal mobile device or a device provided by the study. A research assistant orients participants to the device, provides training on the BCN software, and provides technical support and reminders.
  BCN is a mobile application (app) for informal caregivers of patients with ADRD. The BCN app delivers the following behavioral support:
  1. 24/7 psychoeducation and caregiver support on a variety of ADRD related topics, presented as a browse-able library of stories and advice cards or "Notes";
  2. Assessment of informal caregiver status and patients behavioral and psychological symptoms of dementia (BPSD), in the form of the selfadministered HABC Monitor, along with reporting and historical tracking of HABC Monitor scores;
  3. Engagement tools, in particular, (i) a toolkit for saving, sorting, creating/editing, and sharing Notes and (ii) a bi-directional messaging tool for communicating with clinicians or trusted others.
- Usual Care - Patients: Patients randomized to the comparison group receive usual care for Alzheimer's disease and related dementia (ADRD) from their health system, either Eskenazi Health or Indiana University (IU) Health.
  The standard of ADRD care at Eskenazi Health is the ABC Clinical Program. The goal of the ABC Clinical Program is to help primary care physicians achieve the standard of care in the diagnosis, evaluation and management of patients with ADRD. It is delivered by an interdisciplinary team led by a care coordinator. The informal caregiver of the person living is also enrolled in the program and caregiver burden is assessed and managed. The ABC team collects all relevant data and formulates an individualized care plan in collaboration with the informal caregiver. The care coordinator communicates the team's recommendations to the primary care physician and finalizes a collaborative plan of action. During the next year, the ABC team uses face-to-face and telephone interactions with the patient and caregiver to monitor and modify implementation of the care plan.
  The standard of ADRD care at IU Health is Primary Care visits. The goal of Primary Care at IU Health is to provide preventive care services to their patients. Older adults are assessed for ADRD during clinic visits and referred to brain care specialty as necessary.
- Brain CareNotes (BCN) Software - Patients: Patients randomized to the intervention group continue to receive usual care for ADRD at Eskenazi Health or IU Health, and additionally receive the BCN software.
  BCN is installed on either the caregiver's personal mobile device or a device provided by the study. A research assistant orients participants to the device, provides training on the BCN software, and provides technical support and reminders.
  BCN is a mobile application (app) for informal caregivers of patients with ADRD. The BCN app delivers the following behavioral support:
  1. 24/7 psychoeducation and caregiver support on a variety of ADRD related topics, presented as a browse-able library of stories and advice cards or "Notes";
  2. Assessment of informal caregiver status and patients behavioral and psychological symptoms of dementia (BPSD), in the form of the selfadministered HABC Monitor, along with reporting and historical tracking of HABC Monitor scores;
  3. Engagement tools, in particular, (i) a toolkit for saving, sorting, creating/editing, and sharing Notes and (ii) a bi-directional messaging tool for communicating with clinicians or trusted others.
Arm/Group | Usual Care - Caregivers | Brain CareNotes (BCN) Software - Caregivers | Usual Care - Patients | Brain CareNotes (BCN) Software - Patients
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 1/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/27 | 0/26

LIMITATIONS AND CAVEATS:
BCN usage (a primary feasibility outcome) continues to be analyzed and data are not reported.

Data are reported from consented informal caregivers only. Caregivers provided data on themselves and the patient.

Data on secondary outcomes of Caregiver Burden and Patient Symptom Severity were imputed for all randomized participants.

Acute care utilization data combine emergency room (ER) and hospital based admissions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03119259/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT03119259/ICF_001.pdf